CLINICAL TRIAL: NCT03608202
Title: Impact of a Multisystemic Ultrasound Protocol in Patients of Polyvalent Intensive Care Units. Multicenter Controlled Study
Brief Title: Impact of a Multisystemic Ultrasound Protocol in Patients of Polyvalent Intensive Care Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asociacion Española Primera en Salud (Other)
Collaborators: Intensive Care Unit Pasteur Hospital (Unknown)
Responsible Party: Principal Investigator, Julio Pontet, MD, PhD, Asociacion Española Primera en Salud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AsociacionEPS
Record Dates: First submitted 2017-03-14; First posted 2018-07-31 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Point of Care Ultrasound
Keywords: Intensive Care; Point-of-Care Ultrasound; Thoracic Ultrasound; Diagnostic Techniques and procedures.
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Controlled clinical trial. Prospective, randomized controlled clinical trial. The type of design is with posttest only and control group. Two groups will be compared, a study group ("experimental") undergoing a focal ultrasound protocol, versus a control group with conventional conventional management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POCUS protocol group (Experimental): POCUS protocol group
  It will be submitted to an ultrasound protocol which consists in performing the following ultrasound studies in each patient:
  Measurement of the diameter of the optic nerve. Neck. Pulmonary ultrasound (LUS score). Echocardiogram (function and volemia). Abdomen. Femoral vascular package. Eco-guided interventionism. Central venous accesses (controlling positioning with saline injection under ultrasound), arterial, pleural or abdominal drainage and percutaneous tracheotomy will be performed under ultrasound.
  Interventions: Behavioral: POCUS protocol group
- Control group (Active Comparator): The usual handling will be followed. The studies will only be performed if the medical team-treating team considers it, requesting a radiologist specialist the same, as is done routinely.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: POCUS protocol group — The findings of multiorgan ultrasound can modify diagnoses and treatments and immediate interventions (eg volume loading with saline solution, pleural or pericardial drainage, initiation of diuretics, increase in positive end expiratory pressure, etc.).
  This protocol is performed in the first 24 h of admission to the Intensive Care Unit (ICU) and is repeated at 24 h.
  Arms: POCUS protocol group
Other: Control group — Routine protocol of the treating team is followed
  Arms: Control group

SUMMARY:
Ultrasound is a widely used tool for clinicians to manage severe acute patients, seeking to improve the limitations of traditional physical examination and special studies that require patient transfers and can be harmful. This study aims to determine that a pre-established protocol of multiorganic point-of-care ultrasound can be beneficial performed systematically in a critical care patient, improving the diagnosis, detecting hidden anomalies, generating changes in therapy and guiding interventions. A multicenter, randomized controlled clinical trial, against a conventional therapy group is designed. The study group underwent an ultrasound protocol at the entrance of an ICU, of optic, pulmonary, cardiac, abdominal and guide of interventions.

ELIGIBILITY:
Inclusion Criteria:

• Admitted to the ICU with the requirement of Ventilatory Mechanical Assistance, and admitted for trauma, sepsis, shock of any cause, and postoperative major surgery.

Exclusion Criteria:

* More than 12 hours of previous hospitalization.
* Those who refuse to enter the protocol.
* Those considered by the treating team to be out of recovery possibilities or to enter to support Organ donation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in diagnosis and treatment by point of care ultrasound | Up to 7 days
  REGISTER OF (In terms of frequency):
  IN DIAGNOSIS:
  * Does not modify the initial diagnosis but confirms it
  * Induces a change in initial diagnosis
  * Discover an unknown initial diagnosis
  * Does not modify the initial diagnosis, does not discard or confirm anything and does not change the treatment that is done.
  * Induces a wrong diagnosis and leads to an error.
  IN TREATMENT:
  * Determines the performance of an urgent interventional diagnostic maneuver
  * Determines the performance of an urgent medical or pharmacological therapeutic maneuver of the ICU.
  * Determines the performance of an urgent interventional or surgical therapeutic maneuver

SECONDARY OUTCOMES:
Definitive diagnosis | Up to 7 days
  Delay in performing definitive diagnosis (hours)
ICU extra requirements | Up to 7 days
  Requests for imaging studies (Number per patient)
Interventions | Up to 7 days
  Number and type of procedures or interventions performed on the patient (Number per patient)
Delay times | Up to 7 days
  Delay between the treatment decision and its actual completion (eg pleural drainage) (in hours)
Duration of mechanical ventilation | Up to 30 days
  Time of invasive mechanical ventilation (days)
ICU stay | Up to 30 days
  Internment time in ICU (days)
Mortality | Up to 30 days
  Death rate (percentage)

CONTACTS AND LOCATIONS:
Locations (1):
- UCI Hospital Pasteur y Asociacion Española, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: Yes
Clinical and variable data of multiorganic focal ultrasonography

REFERENCES:
- [Derived] Pontet J, Yic C, Diaz-Gomez JL, Rodriguez P, Sviridenko I, Mendez D, Noveri S, Soca A, Cancela M. Impact of an ultrasound-driven diagnostic protocol at early intensive-care stay: a randomized-controlled trial. Ultrasound J. 2019 Sep 30;11(1):24. doi: 10.1186/s13089-019-0139-2. PMID 31595353